CLINICAL TRIAL: NCT03902431
Title: Implementation Research: Translating the ABCS Into HIV Care
Brief Title: Translating the ABCS Into HIV Care
Acronym: ABCSinHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Clinical Directors Network (Network); University of Texas (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin Fiscella, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: U01HL142107 (NIH); U01HL142107 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV; Cardiovascular Risk Factor

STUDY DESIGN:
Intervention Model Description: A stratified clustered randomized stepped wedge design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): CVD risk prior to the patient and clinician training
- Training (Experimental): CVD risk after the patient and clinician training
  Interventions: Behavioral: ABCS training

INTERVENTIONS:
Behavioral: ABCS training — Clinicians and patients will be given information regarding the ABCS (Aspirin, Blood Pressure control,Cholesterol control, and Smoking Cessation) and for reducing CVD risk among HIV patients.
  Arms: Training

SUMMARY:
The overall objective of this project is to develop and rigorously test implementation strategies to address the gap in scientific knowledge of lower use of evidence-based interventions commonly referred to as the ABCS (aspirin, blood pressure control, cholesterol control, and smoking cessation)which contributes to the growing CVD morbidity and mortality among PLH.

DETAILED DESCRIPTION:
Our project has two major aims:

Aim 1: To assess the impact of the implementation of an evidence-based, multilevel strategy to reduce cardiovascular vascular disease (CVD) among PLH.

Aim 2: To assess the process of implementation of these strategies using RE-AIM QuEST. Using both quantitative and qualitative methods, we evaluate the process of implementation by assessing Reach, [Effectiveness addressed in Aim 1], Adoption, Implementation and Maintenance whilst integrating Qualitative Evaluation for Systematic Translation.

ELIGIBILITY:
Inclusion Criteria:

Sites:

* Serve a cohort of at least 100 HIV patients
* Have an Electronic Health Record (EHR)
* Agree to collaborate on implementing feasible adaptations of intervention strategies

Patients:

* Patient of the site with a diagnosis of HIV
* Age 40-79 years
* ≥5% risk for CVD as calculated using the ASCVD Risk Estimator Plus
* Willing to participate
* No plans to leave the site in the next 12 months
* Proficient in either English or Spanish
* Own a cell phone with texting capabilities

Clinicians:

* Physicians, Physicians Assistants, or Nurse Practitioners who provide direct HIV care to patients
* Work at a participating site
* Willing to implement the project's intervention strategies

Exclusion Criteria:

Patients:

* Currently participating in another CVD trial
* Have experienced a prior cardiac or vascular event such as myocardial infarction (MI) or cerebrovascular accident (CVA)
* Have had a CVD procedure such as installation of a stent or angioplasty
* Have peripheral vascular disease, intermittent claudication or peripheral arterial disease
* Are pregnant
* Lacks capacity to consent

Clinicians:

• Planning to leave the site within the next 12 months

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4277 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
10-year CVD risk reduction | 12 months
  This will be based on the ACVSD risk calculator

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, MD, MPH, Principal Investigator — University of Rochester; Jonathan Tobin, PhD, Principal Investigator — Clinical Directors Network, Inc; Albert Einstein College of Medicine
Locations (1):
- University of Rochester, Rochester, New York, United States